CLINICAL TRIAL: NCT07108140
Title: A Single-Arm, Single-Center, Open-Label Pilot Study of Patients With ALPP-Positive Advanced Solid Tumors
Brief Title: Engineered T-cell Therapy for Patients With ALPP-Positive Advanced Solid Tumors
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Portfolio prioritization
Sponsor: TCRCure Biopharma Ltd. (Industry)
Collaborators: Nanjing University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALPP-NJ002
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: Advanced Solid Tumor; ALPP; CAR-T

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-ALPP CAR-T Cell Therapy (Experimental): Following lymphodepletion chemotherapy, participants will receive anti-ALPP CAR-T cell infusion.
  Interventions: Biological: Anti ALPP CAR-T cells treatment

INTERVENTIONS:
Biological: Anti ALPP CAR-T cells treatment — anti ALPP CAR-T cells Treatment follows a lymphodepletion Drug: Fludarabine and Cyclophosphamide.
  Other Names: Fludarabine Cyclophosphamide

SUMMARY:
This is a single-arm, open-label, dose-escalation clinical trial designed to evaluate the safety, tolerability, expansion, and persistence of ALPP CAR-T cells in patients with ALPP-positive recurrent or metastatic solid tumors who have progressed after prior therapies. The primary objective is to determine the maximum tolerated dose (MTD), with a secondary aim to assess preliminary clinical efficacy in solid tumors.

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label, single-dose clinical trial to evaluate the safety and efficacy of ALPP CAR-T cell therapy in patients with recurrent or metastatic solid tumors. The study protocol consists of five main stages: (1) patient screening, (2) collection of peripheral blood mononuclear cells (PBMCs), (3) lymphodepletion chemotherapy, (4) ALPP CAR-T cell infusion, and (5) post-infusion follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily provide written informed consent.
2. Aged 18-70 years (inclusive).
3. Life expectancy ≥ 3 months.
4. ECOG performance status 0-1.
5. Failed or unsuitable for standard therapy.
6. At least one measurable lesion per RECIST 1.1.
7. ALPP-positive tumor confirmed by immunohistochemistry.
8. Adequate organ and bone marrow function.
9. Effective contraception required for participants of childbearing potential.
10. Adequate venous access for leukapheresis.

Exclusion Criteria:

1. Primary CNS malignancy or uncontrolled CNS metastases.
2. Other malignancies within 5 years (except adequately treated non-melanoma skin cancer or carcinoma in situ).
3. Active autoimmune disease or history of autoimmune disease.
4. Immunodeficiency, including HIV positivity.
5. Bleeding disorders (inherited or acquired).
6. Clinically significant cardiovascular disease.
7. Active infection (including tuberculosis, hepatitis B/C, syphilis).
8. Pregnant or breastfeeding women.
9. History of refractory epilepsy, active GI bleeding, or high risk of tumor bleeding.
10. Severe systemic or psychiatric illness.
11. Prior cell or gene therapy.
12. Severe drug hypersensitivity history.
13. Investigator-assessed unsuitability for trial participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Safety of ALPP CAR-T cells | Up to 24 months
  The incidence, type, and severity of all adverse events, serious adverse events, and abnormal laboratory findings.
Safety of ALPP CAR-T cells | Up to 1 month
  Incidence of DLT

SECONDARY OUTCOMES:
Efficacy of ALPP CAR-T cells | Up to 24 months]
  Optimal objective response rate (ORR)

OTHER OUTCOMES:
To investigate the Cmax of ALPP CAR-T cells in the peripheral blood after infusion | Up to 24 months
To assess ALPP CAR-T cell trafficking into tumor tissues after infusion | Up to 24 months
  To detect ALPP CAR-T cell number in tumor tissues after infusion
To investigate the AUC of ALPP CAR-T cells in the peripheral blood after infusion | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tangfeng Lv, MD, Principal Investigator — The Jinling Hospital
Locations (1):
- The Jinling Hospital, Nanjing, Jiangsu, China